CLINICAL TRIAL: NCT06003023
Title: Establishing Efficacy for the Congenital Heart Disease Physical Activity Lifestyle Intervention
Brief Title: Congenital Heart Disease Physical Activity Lifestyle Study V.2
Acronym: CHD-PALS V2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Jackson (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Jamie Jackson, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002759; R01NR020423 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Heart Defects, Congenital; Cardiovascular Disease Other
Keywords: congenital heart disease; physical activity; adolescents; young adults
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Intervention Model Description: Study includes 2 possible conditions to which participants are randomized: (1) Control: Fitbit + tailored exercise prescription + information on living well with CHD (2) Fitbit + tailored exercise prescription + theory-driven health coaching sessions.
Masking Description: Group assignment will be generated through the data capture system (REDCap) in which the randomization scheme was developed by the study statistician. Investigator, research assistants, coaches (interventionists), and participants do not know which condition a participant is in until after Phase 2 consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Living Well with Congenital Heart Disease (LIV-CHD) Intervention (Active Comparator): In LIV-CHD, participants will receive a Fitbit and a tailored exercise prescription, as devised from their baseline exercise stress test results. They will also meet with a health coach for 9 virtual sessions over a period of 20 weeks. The content will focus on how to use the Fitbit along with health education pertinent to living a healthy lifestyle (e.g., sleep hygiene, stress management). Goal-setting and other cognitive behavioral strategies for health behavior change will not be discussed in this arm. Participants in the attention control arm will also receive text messages reminding them to wear their Fitbit.
  Interventions: Behavioral: Physical Activity Monitoring; Behavioral: Tailored Exercise Prescription; Behavioral: Healthy Lifestyle Education
- Congenital Heart Disease Physical Activity Lifestyle (CHD-PAL) Intervention (Experimental): In CHD-PAL, participants will receive a Fitbit and a tailored exercise prescription, as devised from their baseline exercise stress test results. They will also meet with a health coach for 9 virtual sessions over a period of 20 weeks. The content will focus on cognitive behavioral strategies, grounded in the Theory of Planned Behavior, to increase physical activity and healthy living. Participants in the intervention arm will also receive text motivational messages relevant to session content, as well as reminders to wear their Fitbit.
  Interventions: Behavioral: Physical Activity Monitoring; Behavioral: Tailored Exercise Prescription; Behavioral: Healthy Lifestyle Education; Behavioral: Physical Activity Lifestyle Intervention Informed by the Theory of Planned Behavior

INTERVENTIONS:
Behavioral: Physical Activity Monitoring — A physical activity monitor (Fitbit) will be provided to participants in both arms.
  Other Names: Fitbit
Behavioral: Tailored Exercise Prescription — Participants in both arms will receive the results of their exercise stress test, which includes information on the duration, frequency, and intensity of their physical activity.
Behavioral: Healthy Lifestyle Education — Participants in both arms will receive information on healthy living, including topics such as physical activity, sleep, stress management, and diet.
Behavioral: Physical Activity Lifestyle Intervention Informed by the Theory of Planned Behavior — Participants randomized to the CHD-PAL arm will receive coaching to: 1) change attitudes towards physical activity; 2) increase perceptions of other people's approval of physical activity; 3) increase perceptions of control over being physically active. These elements will be delivered using a non-judgmental stance and will be accompanied by goal-setting.
  Other Names: CHD-PAL
  Arms: Congenital Heart Disease Physical Activity Lifestyle (CHD-PAL) Intervention

SUMMARY:
The Congenital Heart Disease Physical Activity Lifestyle Intervention Study (CHD-PALS) V.2 seeks to determine the efficacy of a lifestyle intervention program for adolescents and young adults (AYAs) with congenital heart disease (CHD). This trial was adapted from the original CHD-PAL trial to continue improving cardiovascular outcomes for transition-aged CHD survivors.

DETAILED DESCRIPTION:
Current estimates indicate more than 2 million individuals in the United States have CHD. CHD survivors are now living well into adulthood, including those with moderate and complex forms of CHD, who previously did not survive childhood. However, adult CHD survivors are now encountering cardiovascular comorbidities, such as coronary disease and hypertension, costing more than $3.16 billion annually in hospitalizations and resulting in premature death. The benefits of physical activity for preventing coronary artery disease and other cardiac comorbidities are well-known. For CHD survivors, the benefits of physical activity for preventing morbidity and premature mortality have also been emphasized. Despite strong evidence for physical activity preventing and treating acquired cardiovascular comorbidities among CHD survivors, adolescents and young adults (AYAs) with CHD do not meet recommended activity levels. The CHD-PAL intervention aims to provide individualized guidance on safe forms of physical activity that is delivered by trained allied health interventionists.

The CHD-PAL intervention is informed by the Theory of Planned Behavior (TPB) which has been used as a framework for lifestyle interventions, including among adults with heart failure and adolescents. Additionally, the CHD-PAL intervention implements goal-setting (or developing action plans) and self-monitoring, both of which are key for enacting the behavior within the TPB.

Investigators will randomize (1:1) 144 AYAs (ages 15-25) with moderate and complex CHD who spend <=30 minutes/day in moderate to vigorous physical activity (MVPA) to 1 of 2 arms: CHD-PAL or attention control (Control). Both arms will receive a Fitbit® and a tailored exercise prescription. Those in CHD-PAL will also receive a 20-week videoconferencing-administered intervention that includes 9, 20 to 30-minute sessions designed to increase positive attitudes towards, subjective norms for, and perceived control for engaging in physical activity. Self-monitoring and goal-setting will also be encouraged to help enact behavior change. Controls will receive the same number/frequency of videoconferencing contacts to discuss the Fitbit and exercise prescription, as well as general healthy living, without addressing the TPB hypothesized mechanisms. Controls will also not be directed to self-monitor or engage in goal-setting. All participants will receive text messages from interventionists to either reinforce session content and inquire about progress towards goals (CHD-PAL) or to remind participants to wear the Fitbit (Control). Randomization will be stratified by gender and age using randomly varying block sizes of 4 to 6. MVPA, as measured with a research-grade accelerometer, will be assessed at baseline (T1), post-intervention (T3; 20 weeks after baseline), interim follow-up (T4; 20 weeks post-intervention), and follow-up (T5; 40 weeks post-intervention). TPB mechanisms will be similarly assessed, with the addition of an interim assessment during the intervention (T2; 10 weeks after baseline). Cardiorespiratory fitness (peak volume of oxygen consumption (VO2) and metabolic equivalent (METs)), as assessed via stress testing, will be measured at T1 and T3 as exploratory secondary outcomes.

The primary aim is to determine the efficacy of the CHD-PAL intervention on change in time spent in moderate to vigorous physical activity (MVPA) for AYAs with moderate and complex CHD. The secondary aim is to explore change in the TPB mechanisms and their relevance to change in MVPA. The tertiary aim is exploring the impact of CHD-PAL on cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-25 years
* Diagnosed with moderate or complex structural CHD
* Actively receiving care from a cardiologist at Nationwide Children's Hospital (NCH) or Ohio State University (OSU)

Exclusion Criteria:

* Unable to speak and read proficiently in English
* Have a diagnosis of a genetic syndrome that impacts multiple organ systems
* Have cognitive impairments that would interfere with completing study measures
* Have been engaged in a formal exercise program within the past 6 months,
* Have participated in the intervention arm of the previous CHD-PAL Study
* Have undergone open-heart surgery or had a valve replacement in the last 3 months
* Are unable to complete an exercise stress test using a treadmill
* Are pregnant
* Are prohibited to engage in at least moderate levels of physical activity by their cardiologist
* Engage in >30 minutes of moderate-to-vigorous physical activity per day, on average per accelerometer
* Have contraindications for exercise based on an exercise stress test (e.g., exercise-induced arrhythmias or evidence of cardiac ischemia)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Moderate to Vigorous Physical Activity (MVPA) | Baseline to Weeks 20, 40, and 80
  Number of minutes spent in moderate to vigorous physical activity as measured by an accelerometer.

SECONDARY OUTCOMES:
Physical Activity Enjoyment/Engagement Scale (Attitudes) | Baseline to Weeks 10, 20, 40, and 80
  18-item measure of enjoyment and dislike of physical activity in which the participant currently engages. Each item is rated on a 7-point Likert scale with a positive attitude (e.g., I enjoy it) and negative attitude (e.g., I hate it) towards physical activity on each end.
Affective Attitudes for Physical Activity Scale (Attitudes) | Baseline to Weeks 10, 20, 40, and 80
  4-item measure of affective physical activity attitudes using bipolar adjectives on a 7-point Likert scale (i.e., enjoyable-unenjoyable, boring-interesting, pleasant-unpleasant, stressful-relaxing).
Physical Activity Norms Measure (Social Norms) | Baseline to Weeks 10, 20, 40, and 80
  5-item measure of perceptions of subjective norms of physical activity (e.g. "Members of my family think I should be physically active regularly"). An additional item was added to assess norms of cardiologist. Original item wording of "during my free time on most days" was changed to "regularly." Participants are presented with a 5-point Likert scale ranging from "Strongly disagree" to "Strongly agree." One item ("Compared to others of your age and sex, mark how active you are.") is measured on a 5-point Likert scale ranging from "Much less active" to "Much more active."
Family and Partner Support for Physical Activity Engagement Measure (Social Norms) | Baseline to Weeks 10, 20, 40, and 80
  39-item measure asking participants to indicate "None," "Rarely," "A few times," Often," "Very often," and "Does not apply," when rating the extent to which family (i.e., parents, siblings) and friends provided support for physical activity in different contexts within the past 3 months. This measure has been modified to include items for partners.
Perceived Control for Physical Activity Engagement Measure (Perceived Control) | Baseline to Weeks 10, 20, 40, and 80
  5-item measure of perceived control for engaging in regular physical activity. Wording was adapted to use "physical activity" instead of "exercise". Each item is rated on a 7-point Likert scale with a negative perception of control (e.g., Very little control) and positive perception of control (e.g., Complete control) of physical activity engagement on each end.
Exercise Confidence Survey (Perceived Control) | Baseline to Weeks 10, 20, 40, and 80
  12-item questionnaire assessing health-related self-efficacy in adjusting physical activity behaviors. The original questionnaire has items for self-efficacy in diet behaviors, which have been removed for the purpose of this study. Wording has also been modified to reflect "physical activity"/"physically active" language. Items are measured on a 5-point Likert scale from "I know I cannot" to "I know I can" with an additional option of "Does not apply."

OTHER OUTCOMES:
Cardiorespiratory Fitness-Volume of Oxygen Consumption (Peak VO2) | Baseline to Week 20
  Peak VO2 is the highest value of oxygen consumption during an exercise stress test and is widely used as an indicator of cardiorespiratory fitness. Peak VO2 will be measured at baseline and post-intervention to examine the impact of CHD-PAL on change in biological markers of cardiovascular health.
Cardiorespiratory Fitness- Metabolic Equivalents (METs) | Baseline to Week 20
  MET scores, or metabolic equivalents, represent the amount of oxygen consumed at rest or during activity. It is a simple, practical way to express the energy cost of different physical activities. METs, as assessed during the exercise stress test, will be measured at baseline and post-intervention to examine the impact of CHD-PAL on change in biological markers of cardiovascular health. METs are calculated by: ([miles per hour x 26.8 x 0.1] + [grade/100 x 1.8 x miles per hour x 26.8] + 3.5)/3.5 and the highest MET achieved during the stress test will be abstracted.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Jackson, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No